CLINICAL TRIAL: NCT00440154
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled,Ezetimibe-Calibrated, Multicenter Study Evaluating the Safety and Efficacy of Four Doses and Two Dose-Regimens of AVE5530 Over 4 Weeks in Patients With Mild to Moderate Primary Hypercholesterolemia
Brief Title: A Study Evaluating the Safety and Efficacy of AVE5530 (4 Weeks) in Patients With Mild to Moderate Hypercholesterolemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRI6589; EudraCT: 2006-005469-20
Record Dates: First submitted 2007-02-23; First posted 2007-02-26 (Estimated); Last update posted 2008-12-16 (Estimated); Status verified 2008-12

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (7):
- 1 (Experimental): oral administration 5 mg breakfast timing
  Interventions: Drug: AVE5530
- 2 (Experimental): oral administration 25 mg breakfast timing
  Interventions: Drug: AVE5530
- 3 (Experimental): oral administration 50 mg breakfast timing
  Interventions: Drug: AVE5530
- 4 (Experimental): oral administration 100 mg breakfast timing
  Interventions: Drug: AVE5530
- 5 (Experimental): oral administration 25 mg dinner timing
  Interventions: Drug: AVE5530
- 6 (Placebo Comparator): oral administration
  Interventions: Drug: placebo
- 7 (Active Comparator): oral administration 10mg breakfast timing
  Interventions: Drug: ezetimibe

INTERVENTIONS:
Drug: AVE5530
  Arms: 1; 2; 3; 4; 5
Drug: placebo
  Arms: 6
Drug: ezetimibe
  Arms: 7

SUMMARY:
The primary objective of this study is to assess the effect of AVE5530 on LDL-C levels over a period of 4 weeks. The secondary objectives are to assess the effects of AVE5530 on other lipid plasma levels and the safety and tolerability of AVE5530.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate primary hypercholesterolemia with stabilized LDL-C baseline ≥130 mg/dL and ≤ 250 mg/dL (≥ 3.36 mmol/L and ≤ 6.46 mmol/L)
* Male aged ≥ 18 years or postmenopausal women at screening

Exclusion Criteria:

* Presence of any clinically significant endocrine disease known to influence serum lipids or lipoproteins
* Patients with type 1 diabetes
* Presence or history of cancer within the past five years
* Triglycerides ≥ 300 mg/dL (3.39 mmol/L)
* Fasting plasma glucose > 160 mg/dL (8.9 mmol/L)
* Impaired kidney function and active liver disease
* Within one month prior to screening visit and/or at the time or after the screening visit, administration of any lipid lowering treatment
* Creatine Kinase > 2xUpper Limit of Normal range

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2007-02; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Percent change in LDL-C from baseline | 4 weeks

SECONDARY OUTCOMES:
Absolute change from in LDL-C levels | 4 weeks
Percent change in other lipids and lipoprotein fractions from baseline | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (6):
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com